CLINICAL TRIAL: NCT04302571
Title: Effects of Home-based Combined Aerobic and Resistance Training on Walking Capacity, Circulating Endothelial Progenitor Cells AND Endothelial Function in Patients With Intermittent Claudication
Brief Title: Effects of Combined Aerobic and Resistance Training in Patients With Intermittent Claudication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Rita Lombardini, Principal Investigator, University Of Perugia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: APE-IC1
Record Dates: First submitted 2020-03-05; First posted 2020-03-10 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Arterial Disease; Endothelial Dysfunction
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy control (No Intervention): Voluntary subjects without peripheral arterial disease
- IC patients, no exercise (Sham Comparator): Patients with peripheral arterial disease stage II (intermittent claudication) on best medical treatment, given advices to perform regular aerobic activity
  Interventions: Behavioral: sham exercise
- IC patients, exercise (Active Comparator): Patients with peripheral arterial disease stage II (intermittent claudication) on best medical treatment, home-based combined physical exercise
  Interventions: Behavioral: combined aerobic and resistance physical activity

INTERVENTIONS:
Behavioral: combined aerobic and resistance physical activity — Five training sessions weekly for 12 weeks are scheduled. Each session lasts 60 minutes divided into 45 minutes of aerobic workout and 15 minutes of circuit training. The aerobic workout consists of walking on a flat floor or on a slight uphill (maximum slope 3%): patients should walk until submaximal walking capacity (80% of their MWT) and rest as they would experience pain at the lower limbs; afterwards, they should start to walk again, once the pain was improved. Resistance training consists of calisthenics exercises focused on trunk and lower limbs muscles (bicycle, flutter kicks, squats, lunges, calf raises, wall sits and power press) with at least 3 repetitions for each exercise, interspersed by 30 seconds recovery. Duration of repetitions increases every 3 weeks.
  Arms: IC patients, exercise
Behavioral: sham exercise — general recommendation to perform regular aerobic physical activity
  Arms: IC patients, no exercise

SUMMARY:
Exercise training improves walking capacity and regional perfusion in patients with Intermittent Claudication (IC). Endothelial Progenitor Cells (EPCs) and Endothelial Microparticles (EMPs) could play an important role in this process, promoting the healing of the diseased endothelium.

The investigators are going to measure EPCs and EMPs in a group of patients with IC and in a control group of healthy individuals before a treadmill test and 2, 24, and 48 hours after the test. Subsequently, a group of IC patients will be randomly assigned to perform a 12-week home-based exercise training program.

The investigators expect a significant increase of EMPs and EPCs after acute and chronic physical activity. We expect also a correlation between the increase of EMPs and EPCs and the improvement in walking capacity. Aim of the study is to demonstrate that acutely performed aerobic exercise could be able to promote the mobilization of EMPs and EPCs in patients with IC and that endothelial progenitor cells mobilization could play a pivotal role in exercise induced improvement of walking performance and endothelial function in subjects with IC.

ELIGIBILITY:
Inclusion Criteria:

* history of stable intermittent claudication (PAD, stage II Fontaine)
* resting ankle-brachial index (ABI) <0,9 and the presence of occlusion or significant stenosis at the color-Doppler duplex ultrasound scanning

Exclusion Criteria:

* lower-limb ischemic rest pain or gangrene (Fontaine stages III and IV)
* inability to obtain the ABI value or to perform a walking test
* exercise tolerance limited by factors other than claudication (i.e., arrhythmias, cardiac symptoms or exaggerated blood pressure rise, severe obesity)
* end-stage liver or renal failure
* acute or chronic inflammatory conditions
* history of recent (<6 months) acute coronary syndrome, cerebrovascular event or inducible myocardial ischemia
* treatment with drugs known to affect walking capacity, including calcium-channel blockers, β-blockers and angiotensin-converting enzyme inhibitors.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Endothelial Microparticles (EMPs) | week 0 - week 12
  hematological parameter, cells particles released by activated endothelium, measured by cytofluorimetry
Endothelial Progenitor Cells (EPCs) | week 0 - week 12
  hematological parameter, immature bone-marrow derived cells which repair the damaged endothelium, measured by cytofluorimetry
Maximum Walking Time | week 0 - week 12
  functional parameter, maximum walking capacity for an individual with IC measured through a treadmill walking test
Pain-free Walking Time | week 0 - week 12
  maximum walking capacity for an individual with IC without experiencing pain measured through a treadmill walking test
Flow-mediated Dilation | week 0 - week 12
  ultrasonographic evaluation of endothelial function

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale "Santa Maria della Misericordia" di Perugia, Perugia, PG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasqualini L, Bagaglia F, Ministrini S, Frangione MR, Leli C, Siepi D, Lombardini R, Marini E, Naeimi Kararoudi M, Piratinskiy A, Pirro M. Effects of structured home-based exercise training on circulating endothelial progenitor cells and endothelial function in patients with intermittent claudication. Vasc Med. 2021 Dec;26(6):633-640. doi: 10.1177/1358863X211020822. Epub 2021 Jun 21. PMID 34151646